CLINICAL TRIAL: NCT03178682
Title: Ultrasound Predictors of Early Pregnancy Failure in Patients With Recurrent Pregnancy Loss
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, lecturer of obstetrics and gynecology, Ain Shams University
Other Study IDs: AinShamsU hospital
Record Dates: First submitted 2017-05-28; First posted 2017-06-07 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Recurrent Pregnancy Loss; Early Pregnancy Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound parameters — ultrasonographic parameters (mean gestational sac diameter, yolk sac diameter, crown rump length, embryonic heart rate and uterine artery Doppler) in predicting early pregnancy failure in patients with recurrent pregnancy loss.

SUMMARY:
evaluation of the role of ultrasonographic parameters (mean gestational sac diameter, yolk sac diameter, crown rump length, embryonic heart rate and uterine artery Doppler) in predicting early pregnancy failure in patients with recurrent pregnancy loss

DETAILED DESCRIPTION:
1. Mean gestational sac diameter (MSD) is determined by measuring the mean of 3 diameters (longitudinal, antero-posterior and transverse) which are measured from inside of the sac excluding the decidual reaction from the measurement. It is normally eccentric in location embedded in endometrium, and has a smooth; round or oval shape.
2. Yolk sac is measured by placing calipers on the inner limits of the longer diameter. It usually appears at the periphery of the gestational sac and should not be floating within the sac. Size of the sac, shape, echogenicity of the rim and center of sac, its number and degenerative changes such as calcification will be evaluated. YS having diameter between 3-7mm, rounded shape, absence of degenerative changes, presence of echogenic rim and hypoechoic center are considered normal. Any deviation from above parameters is considered abnormal.
3. Crown-rump length (CRL) is the length of the embryo from the top of its head to bottom of torso excluding the yolk sac and the extremities, to be measured in sagittal plane of the embryo and recorded as an average of three measurements.
4. The MGSD-CRL ratio was calculated as the difference between the MGSD and the CRL if less than 5 mm are prone to first trimester miscarriage.
5. Embryonic heart rate by M-mode calculated as beat per minute using software of ultrasound machine after measuring by electronic calibers of distance between 2 heart waves on frozen M-mode image.
6. Uterine artery Doppler with measurement of systolic/diastolic (S/D) ratio, resistance index (RI) and pulsatility index (PI) of uterine arteries.

ELIGIBILITY:
Inclusion Criteria:

* A positive pregnancy test result.
* Single intrauterine pregnancy.
* Gestational age by last menstrual period of 6-10 weeks in patients with regular cycles and sure of her last menstrual period date.
* History of recurrent pregnancy loss which is defined as three or more consecutive pregnancy losses.

Exclusion Criteria:

* Women who are uncertain of her last menstrual period date.
* Women with irregular menstrual cycles.
* Multiple pregnancies

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 90 pregnant females with history of recurrent pregnancy loss
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
number of patients develops 1st trimester pregnancy loss | within the first 13 weeks of pregnancy.
  defined as a non-viable intrauterine pregnancy with either empty gestational sac or gestational sac containing embryo or fetus without fetal heart activity

CONTACTS AND LOCATIONS:
Overall Officials: Hassan A Bayomy, MD, Study Director — Professor; Amgad E Abou Gamrah, MD, Study Director — Professor
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided